CLINICAL TRIAL: NCT04355754
Title: Assesment of Usefulness of Ventil Device for Mechanical Ventilation in ICU Patients
Brief Title: Ventil Device Usefulness in Mechanically Ventilated ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Radoslaw Owczuk, full professor, Medical University of Gdansk
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Ventil-COVID-19
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Respiratory Insufficiency
Keywords: critically ill patient; intensive care unit; mechanical ventilation; pandemic
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: The flow divider is connected to the ventilator. Half of the fresh gas flows to the patient, hallf to the artificial lung ( 1:1 ratio). For adequate ventilation tidal volume set on the ventilator is then doubled. Chosen respiratory and circulatory parameters are beeing noted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mechanically ventilated patients (Experimental): Adult ICU patients who are mechanically ventilated and who do not require complex modes of ventilation.
  A designated flow divider (Ventil) will be used to divide inspiratory gas flow from ventilator in two separate streams - one to the patient and the second to the artificial lung
  Interventions: Device: Ventil - a gas flow divider

INTERVENTIONS:
Device: Ventil - a gas flow divider — Checking ventilation parameters set and obtained and clinical parameters while ventilating the patient and an artificial lung simultaneously, using inspiratory flow divider.

SUMMARY:
During Covid-19 pandemic many patients require mechanical ventilation due to disastrous impact of SARS-CoV-2 on lungs. In several countries there is a shortage of ICU beds and ventilators. Critically ill patients are treated outside ICUs. Doctors are facing ethical dilemmas who they should treat with ventilation, who should receive ventilator and who should but will not. In ICUs or step down units or in nursery homes there are also patients beyond hope treated - very often they are dependent on mechanical ventilation. Some attempts to invent a device that could replace complex machines in patients with anticipated poor outcome have been made. Ventil was used in clinical scenarios for separate lung ventilation with good effect. As a flow divider it has a potential to ventilate 2 patients at the same time. In the study Ventil will ventilate one patient and instead of the second there will be an artificial lung. Tidal volumes, minute ventilation, PEEP set and final will be checked. Ppeak, Pmean, Pplat, Cdyn, airway resistance, EtCO2, Sat O2, HR, SAP, DAP will be monitored every 2 hrs, as well as blood-gas analysis (every 8 hrs).

DETAILED DESCRIPTION:
During Covid-19 pandemic many patients require mechanical ventilation due to disastrous impact of SARS-CoV-2 on lungs. In several countries there is a shortage of ICU beds and ventilators. Critically ill patients are treated outside ICUs. Doctors are facing ethical dilemmas who they should treat with ventilation, who should receive ventilator and who should but will not.

Before pandemic in ICUs there had always been patients who required mechanical ventilation because of extrapulmonary reasons as well as palliative cases or those in vegetative condition. Most of these patients require just a simple ventilator, not a sophisticated mode of ventilation. Some attempts to invent a device that could replace complex machines in patients with anticipated poor outcome have been made. Ventil was used in clinical scenarios for separate lung ventilation with good effect. VENTIL device, a flow divider, theoretically allows for independent, fully automated synchronous ventilation of 2 patients with use of only one respirator. In the shortage of respirators (ex. terrorist attack, natural disasters) device allows also to ventilate in classical system two patients using single respirator.

Ventil - independent lung ventilation system was constructed by engineers from Nalecz Institute of Biocybernetics and Biomedical Engineering of Polish Academy of Science. Ventil was tested in the clinical scenario - it's safety had been confirmed. Several years ago the working prototypes of the device, after approval of Ethical Committee, was tested in about 150 patients, who were ventilated with independent synchronous lung ventilation and had been found useful.

The idea of the study is to check the usefulness of the device (modern version) in ICU patients who can be ventilated with volume -controlled mode of ventilation as an attempt to use single device for ventilation of 2 patients. At this moment, according to several scientific societies, sharing mechanical ventilators should not be attempted because it cannot be done safely with current equipment. However, it is possible that using a designed flow divider will allow safe ventilation in patients without needs for complicated modes of ventilation. Then maybe it will be possible to release some ventilators and to use them in patients in severe condition, mainly in the era of extreme ventilator shortage. In the study Ventil will ventilate one patient and instead of the second, there will be an artificial lung. Tidal volumes, minute ventilation, PEEP set and final will be checked. Ppeak, Pmean, Pplat, Cdyn, airway resistance, EtCO2, Sat O2, HR, SAP, DAP will be monitored (every 2 hrs), as well as blood-gas analysis (every 8 hrs)

ELIGIBILITY:
Inclusion Criteria:

* ICU patients who require mechanical ventilation

Exclusion Criteria:

* Patients who require complex modes of ventilation will not be recruited

The sudy in an individual patient be discontinued if case of:

Respiratory Criteria:

* episodes of desaturation <90% (in pts without COPD) without reversibel reason
* need for FiO2 increase by 10%
* need for switch to other than CMV mode of ventillation
* need for neuromucular blockade or for deepen sedation because of assynchrony between patient and venilator
* cummulation of CO2>45 mm Hg (in pts without COPD) not responding to the increase of minute ventilation for 30 minutes
* Pplat >30 cmH2O

Circulatory criteria:

* New haemodynamic disturbances that cannot be explaned by other reasons

  * ↑ or ↓of BP by 20%
  * ↑ or ↓of HR by 20%
  * clinically important heart rhythm disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of cases in which it was necessary to stop using Ventil and to step- back to ventilation without this flow divider | 48 hours
  Ventil will be removed from the patient-ventilator circiuit in case of episodes of desaturation <90% (in pts without COPD) without reversibel reason; need for FiO2 increase by 10%; need for switch to other than CMV mode of ventillation need for neuromucular blockade or for deepen sedation because of assynchrony between patient and venilator cummulation of CO2>45 mm Hg (in pts without COPD) not responding to the increase of minute ventilation for 30 minutes; if Pplat >30 cmH2O; in case of new haemodynamic disturbances that cannot be explaned by other reasons; in case of increase or decrease of BP by 20%; increase or decrease of HR by 20%; in case of occurence of clinically important heart rhythm disturbances

CONTACTS AND LOCATIONS:
Overall Officials: Radoslaw Owczuk, prof, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdansk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided